CLINICAL TRIAL: NCT06291090
Title: In Hospital Treatment of Opioid Use Disorder: Clinician Perspectives and Current Practices
Brief Title: A Multi-site Intervention to Expand Hospital Based OUD Treatment Provision
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-0789; K08DA049905 (NIH)
Record Dates: First submitted 2024-02-20; First posted 2024-03-04 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Opioid Use Disorder
Keywords: opioid use disorder; hospital
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: This intervention will be implemented across 12 hospitals
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- OUD intervention (Experimental): Participants received education on the diagnosis and management of OUD, have access to protocols to walk them through assessment of OUD using Diagnostic and Statistical Manual, fifth Edition (DSM)-5, COWS score to calculate severity of opioid withdrawal, buprenorphine or methadone initiation with pre-populated orders, and clickable links for OUD treatment referral post discharge.
  Interventions: Behavioral: OUD treatment intervention

INTERVENTIONS:
Behavioral: OUD treatment intervention — Participants received education on the diagnosis and management of OUD, have access to protocols to walk them through assessment of OUD using Diagnostic and Statistical Manual, fifth Edition (DSM)-5, COWS score to calculate severity of opioid withdrawal, buprenorphine or methadone initiation with pre-populated orders, and clickable links for OUD treatment referral post discharge.

SUMMARY:
The investigators implemented a multi-site hospital-based opioid use disorder (OUD) treatment intervention across 12 hospitals in Colorado to address an OUD treatment gap among hospitalized adults with OUD.

DETAILED DESCRIPTION:
The investigators implemented a multi-site hospital-based opioid use disorder (OUD) treatment intervention across 12 hospitals in Colorado to address an OUD treatment gap among hospitalized adults with OUD. The intervention included nurse driven universal screening for unhealthy substance use with a social work referral for a brief intervention when indicted, electronic health record-embedded protocols to assess for opioid withdrawal and to direct buprenorphine initiation, methadone orders for opioid withdrawal symptoms, and embedded links for post discharge addiction treatment referral. It also included clinician education and nursing education via video conference or in-person lectures. The intervention was supported by the health system Chief Medical Officer and involved subject matters expertise and representation from nursing leaders, social work leaders, and hospital medicine leaders. Outcomes assess include a pre/post implementation assessment of 1) change in buprenorphine prescribed in hospital and 2) discharge, 3) change in naloxone prescribed, 4) change in hospital based methadone prescribing, and 5) change in average clinical opioid withdrawal scale (COWS) score. investigators also assessed a pre/post survey of hospitalists physicians and advanced practice providers to assess their perception of hospital based OUD treatment provision.

ELIGIBILITY:
Inclusion Criteria:

* Physicians, advanced practice providers, social workers, and nurses who work at any affiliated hospitals

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Change in buprenorphine prescribing at hospital discharge | Calculate monthly prescribing rates over a three year time frame (including pre and post implementation) to assess for change
  Change in rate of buprenorphine prescribing at hospital discharge among patients with OUD before and after intervention implementation

SECONDARY OUTCOMES:
Change in rates of methadone prescribing during hospitalization | Calculate monthly prescribing rates over a three year time frame (including pre and post implementation) to assess for change
  Change in rate of in hospital methadone prescribing among patients with OUD before and after intervention implementation

OTHER OUTCOMES:
Change in average (mean) COWS score over time | Calculate mean monthly COWS scores over a three year time frame (including pre and post implementation) to assess for change
  Change in rate of in mean COWS score among patients with OUD before and after intervention implementation
Change in naloxone prescribing at hospital discharge | Calculate monthly prescribing rates over a three year time frame (including pre and post implementation) to assess for change
  Change in rate of naloxone prescribing at hospital discharge among patients with OUD before and after intervention implementation

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Calcaterra, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medicl Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Calcaterra SL, Lockhart S, Natvig C, Mikulich S. Barriers to initiate buprenorphine and methadone for opioid use disorder treatment with postdischarge treatment linkage. J Hosp Med. 2023 Oct;18(10):896-907. doi: 10.1002/jhm.13193. Epub 2023 Aug 22. PMID 37608527